CLINICAL TRIAL: NCT02743156
Title: Minimizing Contrast Utilization With IVUS Guidance in Coronary Angioplasty to Avoid Acute Nephropathy: The MOZART-II Study
Brief Title: Minimizing Contrast Utilization With IVUS Guidance in Coronary Angioplasty to Avoid Acute Nephropathy
Acronym: Mozart-II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Pedro A. Lemos, Professor of Medicine, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mozart II
Record Dates: First submitted 2016-04-10; First posted 2016-04-19 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Acute Kidney Injury; Acute Renal Failure; Acute Renal Injury
Keywords: IVUS; Acute Renal Failure; Angioplasty; stent; contrast; percutaneous coronary intervention; intravascular ultrasound
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- angiography-guided PCI (Active Comparator): angiography-guided percutaneous coronary intervention
  Interventions: Procedure: Angiography-guided PCI
- IVUS-guided PCI (Experimental): intravascular ultrasound guided percutaneous coronary intervention
  Interventions: Procedure: IVUS-guided PCI

INTERVENTIONS:
Procedure: IVUS-guided PCI — intravascular ultrasound-guided percutaneous coronary intervention
  Other Names: intravascular ultrasound
  Arms: IVUS-guided PCI
Procedure: Angiography-guided PCI — Angiography-guided percutaneous coronary intervention. This is the conventional treatment.
  Arms: angiography-guided PCI

SUMMARY:
Contrast-induced acute kidney injury (CI-AKI) is an important adverse effect of percutaneous coronary interventions. Despite various efforts, very few preventive measures have been shown effective in reducing its incidence.

The final volume of contrast media utilized during the procedure is a well- known independent factor affecting the occurrence of CI-AKI.

Intravascular ultrasound (IVUS) has been largely used as an adjunctive diagnostic tool during percutaneous coronary intervention (PCI). When fully explored, IVUS provides precise information for guiding PCI, thereby reducing the usage of contrast media. Accordingly, the recent MOZART study demonstrated that IVUS may lead to a 2-3-fold decrease in the volume of contrast media during PCI.

In the present study, the hypothesize that IVUS guidance, and its consequent reduction in the volume of contrast media, will in decrease the risk of CI-AKI after PCI, in comparison to standard angiography-guided intervention.

DETAILED DESCRIPTION:
* Prospective, unblinded, randomized (1:1), multi-center trial of 300 patients allocated to one of the treatment arms (IVUS-guided PCI or angiography-guided PCI). Aggressive (non-IVUS) strategies to reduce contrast will be used in both study arms
* The study population will be composed of patients with renal dysfunction referred for PCI of one or more coronary vessels, all of them amenable to IVUS imaging
* After discharge, all subjects will be clinically followed-up for 1 year after the index procedure, at the following time-points: 30 and 180 days and 1 year.
* Unless contra-indicated, all patients elective will receive intravenous hydration during 12 hours pre- and 12 hours post-PCI. For patients with acute coronary syndrome, intensive intravenous hydration should be initiated as early as possible. Saline (NaCl 0.9%) infusion is recommended at a dose of 1 ml / kg body weight per hour, 25 and reduced to 0.5 ml/kg/h for those at high risk of volume overload (e.g. reduced left ventricular function or overt heart failure).The use of N-acetylcysteine or sodium bicarbonate will be left to operator discretion.
* Operators will be strongly recommended to follow strict strategies to reduce the total volume of contrast for all patients
* All percutaneous procedures will be performed using non-ionic, low-osmolar or iso-osmolar, iodine-based contrast media
* The study groups will be compared according to the intention-to-treat principle. Categorical variables will be compared by Fisher's exact testing and continuous variables by Student's T testing. Time-dependent events will be estimated by the Kaplan-Meier method and compared by Hazards Cox modeling or log-rank test

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Coronary artery disease referred for percutaneous intervention, with stent implantation, of one or more epicardial vessel.

  ---->All target lesions must be amenable to IVUS imaging, as judged by an experienced interventionalist (lesions not assessable by IVUS at baseline but which are judged to the assessable at any time during the procedure are eligible).
* Baseline calculated creatinine clearance < 60 ml/min/1.73 m2 or baseline creatinine > 1.5 mg/dl
* Ability to sign informed consent and comply with all study procedures

Exclusion Criteria:

* Use of > 50 ml (single-lesion PCI) or > 70 ml (multi-lesion PCI) of iodinated agents < 72 hours (this restriction includes the contrast used during the diagnostic phase of ad hoc PCI).
* Planned use of iodinated contrast within the next 72 hours after the index procedure
* Use of other nephrotoxic agents < 7 days
* Known allergy to contrast agents
* Unstable or unknown renal function prior to PCI.
* Prior PCI of the target lesions
* Patients requiring additional surgery (cardiac or non cardiac) within 72 hours after the index procedure
* Non cardiac co-morbidities with life expectancy less than 1 year
* Other investigational drug or device studies that have not reached their primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Contrast-induced acute kidney injury | 72 hours
  Evaluate whether IVUS-guided PCI reduces CI-AKI in
  comparison to stand-alone angiography-guided PCI. CI-AKI will be defined as
  an increase in serum creatinine ≥ 0.5 mg/dl from the baseline value, within
  72 hours after the index procedure (or at discharge).

SECONDARY OUTCOMES:
Major adverse cardiac events and components | one year
  cardiovascular death, myocardial infarction and target vessel revascularization
Stent thrombosis | one year
  stent thrombosis will be defined as the occurrence of definite or probable stent thrombosis according to the Academic Research Consortium (ARC) criteria
Serious acute kidney dysfunction | one year
  increase in serum creatinine ≥ 2 mg/dl or need for dialysis
Procedure Time | procedure time
Radiation exposure | procedure time

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A. Lemos, MD PhD, Principal Investigator — Heart Institute - InCor. University of Sao Paulo Medical School
Locations (2):
- Heart Institute - InCor. University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil
- Hospital Clinic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided